CLINICAL TRIAL: NCT03615586
Title: The Use of Chaperone in Routine First Visit Anorectal Examination of Women
Brief Title: The Use of Chaperone in Routine Anorectal Examination
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 17-0597
Record Dates: First submitted 2018-07-30; First posted 2018-08-06 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-07

CONDITIONS: Exanimation
MeSH Terms: conditions — Coma | interventions — Molecular Chaperones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With Chaperone (Active Comparator): Female patients examined by male physicians in the presence of a female (nurse) chaperone. The intervention consists of the presence of a female chaperone.
  Interventions: Other: With Chaperone
- Without Chaperone (Active Comparator): Female patients examined by male physicians without a chaperone. The intervention is the absence of a female chaperone.
  Interventions: Other: Without Chaperone

INTERVENTIONS:
Other: With Chaperone — Female patients examined by male physicians in the presence of a female (nurse) chaperone.
  Arms: With Chaperone
Other: Without Chaperone — Female patients examined by male physicians without the presence of a female (nurse) chaperone.
  Arms: Without Chaperone

SUMMARY:
Background and aim: The use of chaperone in routine anorectal examination of women attending to Coloproctology clinics has not been studied to this date. The aim of this study is to compare the patients' perception and preference regarding the presence of a chaperone during their first anorectal examination. Patients and methods: adult women will be randomly selected to be examined with or without the presence of a female chaperone. After that, they will answer a questionnaire form about how they feel during the examination and whether or not they would prefer having or not a chaperone present in that clinical situation. The patients will prospectively enrolled in one of the two groups of this randomized trial during a period of two years.

DETAILED DESCRIPTION:
The use of chaperone in routine anorectal examination of women attending to Coloproctology clinics has not been studied to this date. However, there are some guidance saying says that doctors should offer the patient the option of a chaperone wherever possible before conducting an intimate examination. The aim of this study is to compare the female patients' perception and preference regarding the presence of a chaperone during their first anorectal examination conduct by a male physician. Adult women will be investigated during their first visit to a Coloproctology Clinic at University Hospital. Only senior professionals will be examining the patients. This will be a prospectively randomized trial. Patients will be selected to be examined with or without the presence of a female chaperone. After that, they will answer a questionnaire form about how they feel during the examination and whether or not they would prefer having or not a chaperone present during the anorectal examination. The enrollment period will be two years from July 2018. Sample size estimated for the study is 188 patients (94 in each study group).

ELIGIBILITY:
Inclusion Criteria:

* adult female patients;
* first visit to our Coloproctology clinic;
* signed consent form

Exclusion Criteria:

* patients previously submitted to anorectal examination;
* refusal of participation.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female patients can be eligible for the study
Enrollment: 188 (Estimated)
Dates: Start 2018-07-26 (Actual); Primary Completion 2020-07-26 (Estimated); Study Completion 2020-07-27 (Estimated)

PRIMARY OUTCOMES:
Preference to have or not chaperone during anorectal examination. | Only one assessment by a questionnaire right at the end of clinical visit (1 minute after completing the visit).
  Assessed by the question: "Would you rather have taken the exam in the (without) presence of another person (woman)?". There are 3 possible answers: yes, no, indifferent.

SECONDARY OUTCOMES:
Degree of comfort during anorectal examination. | Only one assessment by a questionnaire right at the end of clinical visit (1 minute after completing the visit).
  Assessed by a specific question: "How did you feel during the exam?" Patients will register their answer in a scale from zero (completely embarrassed) to 10 (completely confortable)
Patients's feeling about having or not chaperone during anorectal examination. | Only one assessment by a questionnaire right at the end of clinical visit (1 minute after completing the visit).
  Assessed by the question: "What did you think of (not) having a person besides the doctor during the exam?" Patients will have 3 possible answers: bad, indifferent, good.
Evaluation of the anorectal examination according to the presence or absence of a chaperone | Only one assessment by a questionnaire right at the end of clinical visit (1 minute after completing the visit).
  Question: "Do you think the (absence) presence of another person made the examination" . There are 3 possible answers: better, worse, did not change it.
Feeling of protection during anorectal examination according to the presence or absence of a chaperone | Only one assessment by a questionnaire right at the end of clinical visit (1 minute after completing the visit).
  Question: "Did you feel more (less) protected with (without) the presence of another person?" There are 3 possible answers: yes, no, indifferent.
Preference to have a chaperone in a future anorectal examination | Only one assessment by a questionnaire right at the end of clinical visit (1 minute after completing the visit).
  Question: "In the event of a reexamination, would you want another person's presence again?" There are 3 possible answers: yes, no, indifferent.
  Or: "Would you again like the doctor to examine you without another person's presence?" There are 3 possible answers: yes, no, indifferent.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C Damin, MD, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gawande A. Naked. N Engl J Med. 2005 Aug 18;353(7):645-8. doi: 10.1056/NEJMp058120. No abstract available. PMID 16107618
- [Background] Stagno SJ, Forster H, Belinson J. Medical and osteopathic boards' positions on chaperones during gynecologic examinations. Obstet Gynecol. 1999 Sep;94(3):352-4. doi: 10.1016/s0029-7844(99)00301-4. PMID 10472858
- [Background] Ehrenthal DB, Farber NJ, Collier VU, Aboff BM. Chaperone use by residents during pelvic, breast, testicular, and rectal exams. J Gen Intern Med. 2000 Aug;15(8):573-6. doi: 10.1046/j.1525-1497.2000.10006.x. PMID 10940150
- [Background] Conway S, Harvey I. Use and offering of chaperones by general practitioners: postal questionnaire survey in Norfolk. BMJ. 2005 Jan 29;330(7485):235-6. doi: 10.1136/bmj.38320.472986.8F. Epub 2004 Dec 16. No abstract available. PMID 15604154
- [Background] Whitford DL, Karim M, Thompson G. Attitudes of patients towards the use of chaperones in primary care. Br J Gen Pract. 2001 May;51(466):381-3. PMID 11360703
- [Background] Teague R, Newton D, Fairley CK, Hocking J, Pitts M, Bradshaw C, Chen M. The differing views of male and female patients toward chaperones for genital examinations in a sexual health setting. Sex Transm Dis. 2007 Dec;34(12):1004-7. doi: 10.1097/OLQ.0b013e3180ca8f3a. PMID 17621250
- [Derived] Damin DC, Contu PC, Savaris RF, Biazi B. Women's preferences regarding the use of chaperones during proctological examinations conducted by male physicians: a randomised clinical trial. Int J Colorectal Dis. 2025 Jan 2;40(1):3. doi: 10.1007/s00384-024-04796-4. PMID 39745520

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-05): https://cdn.clinicaltrials.gov/large-docs/86/NCT03615586/Prot_SAP_001.pdf